CLINICAL TRIAL: NCT04305418
Title: The Efficacy of Mindfulness- Based Intervention for Systemic Lupus Erythematosus (SLE): a Randomized Control Trial
Brief Title: Mindfulness- Based Intervention for Systemic Lupus Erythematosus (SLE) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bar-Ilan University, Israel (Other)
Responsible Party: Principal Investigator, Danny Horesh, Senior lecturer and head of the Trauma and Stress Research Lab at Bar-Ilan University's Department of Psychology., Bar-Ilan University, Israel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25112019
Record Dates: First submitted 2020-02-24; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Psychological
Keywords: Mindfulness; MBSR; Systemic Lupus Erythematosus (SLE); Rheumatic disease; Psychological Stress
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Rheumatic Diseases; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: The current study is a randomized- Control Trial (RCT), 26 patients diagnosed with Systemic Lupus Erythematosus (SLE) were randomly assigned either to mindfulness-based intervention group (MBI) or to a wait-list control group (WL).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, therapists and outcome assesors are blind to the condition the individual participant was assigned to, by encrypting the names of the individual into a number-letter codes.
  The therapists led the intervention group was not aware of the participants condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness- Based Intervention (MBI) (Experimental): In MBI arm, patients received mindfulness- based intervention, a psychological mind- body intervention, focusing on stress reduction,. the intervention was led by a licensed clinical therapist and mindfulness specialist, who was trained in MBSR at Bangor University.
  Interventions: Other: Mindfulness- Based Intervention
- Wait- List Controls (WL) (No Intervention): Patients in wait- list control arm received no active treatment during their 10-weeks waiting period. At the end of that period received the exact intervention as the study group.

INTERVENTIONS:
Other: Mindfulness- Based Intervention — Mindfulness- Based Intervention in a psychological intervention, based on mind- body connection.
  The protocol includes a 10- weeks program, with weekly group sessions of 2 hours and one all-day session after seven weeks. The intervention have standardized core elements consisting of different mental and physical mindfulness exercises: 1) body-scan exercises (paying close attention to all body parts, from the feet to the head), 2) mental exercises focusing one's attention on breathing, 3) physical exercises with focus on being aware of bodily sensations and one's own limits during the exercises, and 4) practicing being fully aware during everyday activities by using the breath as an anchor for attention. Essential to all parts of the program is developing an accepting and non-reactive attitude to what one experiences in each moment.
  Arms: Mindfulness- Based Intervention (MBI)

SUMMARY:
Systemic lupus erythematosus (SLE) is a rheumatic autoimmune disease, involving chronic pain, fatigue, movement difficulties, and is often accompanied by tremendous psychological and psychiatric difficulties. Mindfulness-based Intervention (MBI), is a mind-body intervention, which has been documented in several studies as effective among stress- related diseases, such as crohn's disease.

Nevertheless, not much is known about the efficiency of MBI among SLE patients and about the mechanisms of change through which MBI works. In the present study, the investigators are focusing on different cognitive mechanisms and their role in MBI action.

The study is a randomized-controlled trial. 26 Patients diagnosed with SLE (Mean age=41.26) were randomly assigned to either a 10-weeks MBI intervention (N=15) or a waitlist-control (WL;N=11).4 central measurements points were conducted through the study, which included physiological and psychological variables: at the beginning of the intervention (T1), in the middle of the intervention (T2) at the end of the intervention (T3) and one 6 months follow- up measurement after the termination of the intervention (T4). additionally, participant's blood test has been taken at the beginning and at the end of the intervention.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) Systemic lupus erythematosus (SLE) is an inflammatory autoimmune disease, fluctuates between mild to severe, involving chronic fatigue, Joint pain, stiffness and swelling, often display skin lesions that appear or worsen with sun exposure.

SLE is a stress-related disease, and in many cases, symptoms are worsened under stressful conditions. Studies which have examined the role of stress in maintaining and exacerbate of the disease, have found a large impact of daily stress on the severity of joint pain, abdominal distress, and rash.

Lupus has a high comorbidity with psychiatric disorders. Throughout their lives, 65% of patients with lupus are diagnosed with a mood or anxiety disorder, including major depression (47%), specific phobia (24%), panic disorder (16%), obsessive-compulsive disorder (9%), and bipolar disorder.

Mindfulness Mindfulness involves 'paying attention in a particular way: on purpose, in the present moment, and nonjudgmentally'. It refers to the cultivation of conscious awareness and attention on a moment-to-moment basis. The quality of awareness sought by mindfulness practice includes openness or receptiveness, curiosity and a non-judgmental attitude. An emphasis is placed on seeing and accepting things as they are without trying to change them. With its emphasis on acceptance of body sensations, it should come as no surprise that mindfulness was found to be effective in treating a variety of medical conditions, where distress often stems from the intrusive nature of the pain and difficulties in daily functioning Mindfulness-based stress reduction (MBSR) MBSR is a mindfulness based intervention, developed at the University of Massachusetts Medical Center in 1979 as an intervention to relieve stress and better cope with illness, and it is now being offered at many health care institutions in the US and Europe. In its original version, MBSR is an eight-week program in mindfulness training. The standard program has weekly group sessions of 2 - 2.5 hours and one all-day session after six to seven weeks. The weekly sessions have standardized core elements consisting of different mental and physical mindfulness exercises: 1) body-scan exercises (paying close attention to all body parts, from the feet to the head), 2) mental exercises focusing one's attention on breathing, 3) physical exercises with focus on being aware of bodily sensations and one's own limits during the exercises, and 4) practicing being fully aware during everyday activities by using the breath as an anchor for attention. Essential to all parts of the program is developing an accepting and non-reactive attitude to what one experiences in each moment.

MBSR interventions have never been studied among patients with SLE, and this study is the first randomized- controlled trial which explore the efficacy of mindfulness- based intervention among SLE patients. Additionally, Recent years have seen a surge in research supporting personalized treatment, "tailored" to the individual patient's size. Various studies have shown a significant interaction between specific patient characteristics and treatment outcome. Nonetheless, most research in the field of Mindfulness have used the standard protocol of MBSR, without considering the specific need and difficulties of SLE patient, both psychological and physical (e.g., sitting down through a long meditation). In the current study, the investigators plan to answer this gap, and develop a protocol of MBI (mindfulness- based intervention) based on the generic MBSR protocol, which would be adapted to the specific needs of SLE patients.

The main objective of this study is to explore the impact of MBI on SLE patients. Since SLE is a stress-related conditions, which is maintained and worsened by stress, the investigators believe that an intervention which focuses on stress- reduction, such as MBI, would be very beneficial for the condition, and that the reduction in stress would mediate an improvement in physiological aspects (e.g., pain), psychological aspects (e.g., depression and anxiety) and cognitive aspects (e.g., control of pain and body awareness) of the conditions as well.

Recent years have seen a surge in research supporting personalized treatment, "tailored" to the individual patient's size. Various studies have shown a significant interaction between specific patient characteristics and treatment outcome.

In this study, the investigators will examine how potential cognitive (e.g., psychological flexibility towards pain, pain catasrophizing), psychopathological (e.g., baseline stress and depression) and physiological (e.g., baseline Lupus symptoms) moderators of MBI action.

In this study, for the first time ever, the investigators explore an amended MBSR protocol, which has been tailored specifically to address the unique and exclusive necessities and adversities of SLE patients, such as pain and the cognitive psychological aspects of the pain. This examination is highly supported by the approach of personalized medicine, which has significantly developed over the last decades, advocating the creation of customized treatment, which is "tailored" to the patient's size.

the investigators expect that MBI would lead to greater improvements in clinical symptoms (such as depression and anxiety), decrease pain levels and enhance cognitive processes such as psychological flexibility, compared to a waiting list control group.

Consequently, the investigators assume that the expected reduction in symptoms, would be mediated by cognitive variables, namely, a positive change in cognitive variable, in turn, will lead to positive changes in psychological and physiological symptoms.

Methods The current study is a randomized- Control Trial (RCT), 119 patients diagnosed with SLE syndrome were randomly assigned either to mindfulness-based intervention group (MBI) or to a wait-list control group (WL).

MBI group Treatment participants received MBI, specially adapted to treat SLE patients by a group of mindfulness specialist psychologists and therapists. The intervention led by a licensed clinical therapist and mindfulness specialist, who was trained in MBSR at Bangor University.

The intervention took place in Chaim Sheba medical Center and lasted 10 weeks, with one session a week.

the investigators conducted 4 central measurements points through the study, which included physiological and psychological variables: at the beginning of the intervention (T1), in the middle of the intervention (T2) at the end of the intervention (T3) and one 6 months follow- up measurement after the termination of the intervention (T4). Additionally, the investigators conducted blood tests before and after the intervention (T1 and T3).

In addition to the quantitative date, the investigators carried out qualitative interviews, in order to examine the experience of the participants in the intervention in their own words. The aims of the interviews were to explore participants' subjective experiences in their own words, to acquire a deeper understand of the changes in psychological aspects and to analyze the underlying mechanisms of psychological changes. Furthermore, the investigators wanted to comprehend the specific needs of SLE patients might be better addressed within the adapted protocol.

Last, blood tests were conducted before and after the intervention (T1 and T3), in order to examine blood related measures, including a c-reactive protein test (CRP), erythrocyte sedimentation rate, complement C3 and C4, cytokines, antibodies and Complete Blood Count (CBC).

Wait-list control group Patients randomized to this group received no active treatment during their 10-weeks waiting period, and in the end of that period received the exact intervention as the study group.

ELIGIBILITY:
Inclusion Criteria:

1. confirmation of a clinical diagnosis of Lupus by the patient's own physician
2. age 18 years or older
3. Hebrew speakers
4. physical ability to attend group intervention sessions
5. psychological ability to practice mindfulness (no cognitive extreme impairments, no psychosis, no suicidal tendencies)

Exclusion Criteria:

1. serious mental health condition (such as suicidal state, alcohol and drug abuse, schizophrenia)
2. serious physical condition that would not enable participation
3. participation in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-08 (Actual)

PRIMARY OUTCOMES:
Systemic Lupus Activity Questionnaire | Through study completion, an average of 9 month
  Systemic Lupus Activity Questionnaire (SLAQ), to assess self-reported lupus activity . An analog to the Systemic Lupus Activity Measure (SLAM), the SLAQ includes 24 questions related to disease activity in SLE. Items are weighted and aggregated in a manner analogous to the scoring system used in the SLAM, and scores range from 0-44, with higher scores indicating greater disease activity. The SLAQ is highly correlated with physicians' ratings of disease activity, and other health indices, including the Short Form 12 Health Survey physical component summary and the Short Form 36 physical functioning subscale.
PSS (Perceived Stress Scale) | Through study completion, an average of 9 month
  A widely-used and well-validated 10-item scale that measures the degree to which situations in one's life over the past month are appraised as unpredictable, uncontrollable and overwhelming. It posits that people appraise potentially threatening or challenging events in relation to their available coping resources. Items are rated on a Likert scale ranging from 0 (never) to 4 (very often). A higher score indicates a greater degree of perceived stress. The PSS was often found to possess very good psychometric properties.
PHQ-9 (The Patient Health Questionnaire-9 ) | Through study completion, an average of 9 month
  PHQ-9 is a self-administered questionnaire used to assess major depression symptoms, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). It can yield either a continuous score, or a probable major depressive disorder diagnosis using a cut-off of 10. The sensitivity and specificity of the PHQ-9 compare favorably with structured psychiatric interviews and the Cronbach alpha was found to be 0.89 in a sample of primary care patients.
FFMQ (Five Facet Mindfulness Questionnaire) | Through study completion, an average of 9 month
  FFMQ derived from a factor analysis of questionnaires measuring a trait-like general tendency to be mindful in daily life. It yield five scoring scales that appear to represent elements of mindfulness as it is currently conceptualized: observing, describing, acting with awareness, non-judging of inner experience, and non- reactivity to inner experience. FFMQ consists of 39 items, items are rated on a Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true). The FFMQ has been shown to have good internal consistency and significant relationships in the predicted directions with a variety of constructs related to mindfulness.
PIPS (Psychological Inflexibility in Pain Scale) | Through study completion, an average of 9 month
  PIPS is a 12-item scale developed to assess target variables in exposure and acceptance-oriented treatments of chronic pain ("I postpone things because of my pain"). The subscales measure avoidance (eight items) and cognitive fusion (four items). Items can be answered on a 7-point Likert scale (1=never true to 7=always true). The total score ranges from 12 to 84 points. Higher scores indicate greater psychological inflexibility. Studies showed good model fit and internal consistencies.
PCS (The pain catastrophizing scale) | Through study completion, an average of 9 month
  The PCS is a self-administered questionnaire that consists of 13 items to assess the extent of the patient's catastrophizing thoughts and behaviors. It comprises three subscales: helplessness, magnification, and rumination. The questionnaire is completed in relation to the patient's thoughts and feelings when they are in pain. The scores for the subscales are given by the sum of the corresponding items, and the total score is computed by summation of all items. The PCS score ranges from 0 to 52 points.
EQ (Experiences Questionnaire) | Through study completion, an average of 9 month
  EQ is a 20-item self-report scale measuring decentering, in which participants rate items on a 7-point Likert-type scale (1 = never to 7 = all the time). It evaluates an individual's ability to decenter, namely, the ability to regard thoughts and feelings as temporary and transient. The EQ focuses on three facets of decentering: the ability to view one's self as separate from one's thoughts, the ability to non-judgmentally observe one's negative experiences without habitually reacting, and the capacity for self-compassion. Multiple studies have demonstrated sound psychometric properties of the EQ.
BAI (The Beck Anxiety Inventory) | Through study completion, an average of 9 month
  BAI is a 21-item questionnaire that measures cognitive and somatic symptoms of anxiety, with higher scores indicating increased anxiety, (range 0-63). Sample items include "unable to relax" and "heart pounding or racing." Good psychometric properties have been demonstrated among college, medical, and psychiatric samples. The BAI is a 21-item scale that measures cognitive, somatic, and affective symptoms of anxiety.
BAQ (Body awareness questionnaire) | Through study completion, an average of 9 month
  The 18-item Body Awareness Questionnaire assessed reported attentiveness to normal non-emotive body processes, sensitivity to body cycles/rhythms, ability to detect small changes in normal functioning, and to anticipate bodily reactions ("I am aware of a cycle in my activity level throughout the day", and "I notice specific bodily reactions to being over hungry"). It is a 7-point Likert-type scale (1 = Not at all true of me to 7 = Very true of me). Studies reported good reliability and validity of the BAQ. The total score ranges from 18 to 126 points. Higher scores indicate greater body awareness.
The WHOQOL-BREF (The World Health Organization Quality of Life) | Through study completion, an average of 9 month
  WHOQOL is an abbreviated 26-item version of the WHOQOL-100, on a scale of 1-5. It contains one general QOL item, one general health item, and 24 specific items-one item from each of the 24 QOL facets of the WHOQOL-100. The 24 specific items cover four broad domains: physical, psychological, social, and environmental quality of life. The items are answered on five-point scales, which assess the intensity, capacity, frequency, and evaluation of QOL facets with respect to the last two weeks. Negatively keyed items are reversely scored, so that higher values indicate better QOL.
VAS Pain (Visual Analog Scale for Pain) | Through study completion, an average of 9 month
  The VAS pain is a self- report measure continuous scale, comprised of a horizontal line ranged of 0-100. VAS was based on 3 single- item continuous scale, for pain intensity, shame in one's disease and the third measured the levels of how much the disease has taken over the patients identity. The VAS is the most commonly used measure for assessing levels of pain by physicians in medical setting.
DAI-10 (Drug Attitude Inventory) | Through study completion, an average of 9 month
  The DAI includes a series of 10 questions, each with true/false answers, regarding the adherent of patients to their prescribed medication, and pertaining to various aspects of the patient's perceptions and experiences of treatment. The original scale consists of 30 questions, but a short form consisting of 10 questions has also been validated.
Home Practice Diary | Through study completion, an average of 9 month
  In order to comprehensively assess mindfulness practice at home, participants would fill out a daily home practice diary, which will include the date, time, type, and duration of both formal and informal mindfulness home practice, along with any comments on their experience. This home practice form is commonly used in MBSR interventions.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Chaim Sheba Medical Center, Ramat Gan
  - Bar- Ilan University, Ramat Gan

IPD SHARING:
Plan to Share IPD: Yes
IPD would be available to other researchers, including Study Protocol, Statistical Analysis Plan, Informed Consent Form, Clinical Study Report and Analytic Code through e- mail or publications.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Adams SG Jr, Dammers PM, Saia TL, Brantley PJ, Gaydos GR. Stress, depression, and anxiety predict average symptom severity and daily symptom fluctuation in systemic lupus erythematosus. J Behav Med. 1994 Oct;17(5):459-77. doi: 10.1007/BF01857920. PMID 7877156
- [Background] Cervera R, Khamashta MA, Font J, Sebastiani GD, Gil A, Lavilla P, Mejia JC, Aydintug AO, Chwalinska-Sadowska H, de Ramon E, Fernandez-Nebro A, Galeazzi M, Valen M, Mathieu A, Houssiau F, Caro N, Alba P, Ramos-Casals M, Ingelmo M, Hughes GR; European Working Party on Systemic Lupus Erythematosus. Morbidity and mortality in systemic lupus erythematosus during a 10-year period: a comparison of early and late manifestations in a cohort of 1,000 patients. Medicine (Baltimore). 2003 Sep;82(5):299-308. doi: 10.1097/01.md.0000091181.93122.55. PMID 14530779
- [Background] Emmelkamp, P. M., Bouman, T. K., & Blaauw, E. (1994). Individualized versus standardized therapy: A comparative evaluation with obsessive-compulsive patients. Clinical Psychology & Psychotherapy, 1(2), 95-100.
- [Background] Emori A, Matsushima E, Aihara O, Ohta K, Koike R, Miyasaka N, Kato M. Cognitive dysfunction in systemic lupus erythematosus. Psychiatry Clin Neurosci. 2005 Oct;59(5):584-9. doi: 10.1111/j.1440-1819.2005.01418.x. PMID 16194262
- [Background] Glass JM. Review of cognitive dysfunction in fibromyalgia: a convergence on working memory and attentional control impairments. Rheum Dis Clin North Am. 2009 May;35(2):299-311. doi: 10.1016/j.rdc.2009.06.002. PMID 19647144
- [Background] Hamburg MA, Collins FS. The path to personalized medicine. N Engl J Med. 2010 Jul 22;363(4):301-4. doi: 10.1056/NEJMp1006304. Epub 2010 Jun 15. No abstract available. PMID 20551152
- [Background] Kazdin AE. Understanding how and why psychotherapy leads to change. Psychother Res. 2009 Jul;19(4-5):418-28. doi: 10.1080/10503300802448899. PMID 19034715
- [Background] Kabat-Zinn J. An outpatient program in behavioral medicine for chronic pain patients based on the practice of mindfulness meditation: theoretical considerations and preliminary results. Gen Hosp Psychiatry. 1982 Apr;4(1):33-47. doi: 10.1016/0163-8343(82)90026-3. PMID 7042457
- [Background] Kabat-Zinn J, Lipworth L, Burney R. The clinical use of mindfulness meditation for the self-regulation of chronic pain. J Behav Med. 1985 Jun;8(2):163-90. doi: 10.1007/BF00845519. PMID 3897551
- [Background] Karlson EW, Daltroy LH, Rivest C, Ramsey-Goldman R, Wright EA, Partridge AJ, Liang MH, Fortin PR. Validation of a Systemic Lupus Activity Questionnaire (SLAQ) for population studies. Lupus. 2003;12(4):280-6. doi: 10.1191/0961203303lu332oa. PMID 12729051
- [Background] Liang MH, Socher SA, Larson MG, Schur PH. Reliability and validity of six systems for the clinical assessment of disease activity in systemic lupus erythematosus. Arthritis Rheum. 1989 Sep;32(9):1107-18. doi: 10.1002/anr.1780320909. PMID 2775320
- [Background] Meszaros ZS, Perl A, Faraone SV. Psychiatric symptoms in systemic lupus erythematosus: a systematic review. J Clin Psychiatry. 2012 Jul;73(7):993-1001. doi: 10.4088/JCP.11r07425. Epub 2012 May 1. PMID 22687742
- [Background] Morone NE, Greco CM, Weiner DK. Mindfulness meditation for the treatment of chronic low back pain in older adults: a randomized controlled pilot study. Pain. 2008 Feb;134(3):310-319. doi: 10.1016/j.pain.2007.04.038. Epub 2007 Jun 1. PMID 17544212
- [Background] Schulte, D., Künzel, R., Pepping, G., & Schulte-Bahrenberg, T. (1992). Tailor-made versus standardized therapy of phobic patients. Advances in Behaviour Research and Therapy, 14(2), 67-92.
- [Background] Yazdany J, Yelin EH, Panopalis P, Trupin L, Julian L, Katz PP. Validation of the systemic lupus erythematosus activity questionnaire in a large observational cohort. Arthritis Rheum. 2008 Jan 15;59(1):136-43. doi: 10.1002/art.23238. PMID 18163398
- [Background] Wallace DJ. The role of stress and trauma in rheumatoid arthritis and systemic lupus erythematosus. Semin Arthritis Rheum. 1987 Feb;16(3):153-7. doi: 10.1016/0049-0172(87)90018-7. PMID 3547654